CLINICAL TRIAL: NCT03890315
Title: Evaluation of Patients With Neuropathic Pain in the Context of Clinical Symptoms, Quantitative Sensory Tests and Imaging With FMRI
Brief Title: Evaluation of Neuropathic Pain in the Context of Clinical Symptoms, Quantitative Sensory Tests and Imaging With FMRI
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Göksel Tanıgör M.D., Researcher, Ege University
Other Study IDs: QST-FMRI
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Neuropathic Pain; Radiculopathy, Cervical
MeSH Terms: conditions — Neuralgia; Radiculopathy | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuropathic pain: Adult patients with upper extremity neuropathic pain due to radiculopathy Duration of >1 month Unilateral extremity pain will be recruited
  Interventions: Diagnostic Test: Functional MRI
- Control: Age and gender matched control patients will also be recruited to show whether differences exist in outcome measures.
  Interventions: Diagnostic Test: Functional MRI

INTERVENTIONS:
Diagnostic Test: Functional MRI — In fMRI, patients will first be taking a resting state phase in case of activations. In the block design phase, they will be given tactile stimuli in affected extremity, and then healthy extremity in 3 blocks, followed by pauses.
  Primary and secondary sensorial cortex, insular cortex, anterior cingulate cortex, preforntal cortex and amygdala activation will be chosen as regions of interest, and their activation will be recorded for analyses.

SUMMARY:
This study is planned to evaluate patients with upper extremity neuropathic pain due to cervical radiculopathy with clinical symptoms, Quantitative Sensory Testing(QST) and Functional Magnetic Resonance Imaging(fMRI). Patients with similar charactheristics will be grouped and comparisons will be conducted in fMRI results, as well as QST.

DETAILED DESCRIPTION:
Neuropathic pain is a type of pain which usually accompanies injuries or conduction defects in the central or peripheral nervous system, as well as receptors. Unlike the other types of pain, neuropathic ones are more resistant to therapy and prone to be chronic.

In recent years, there are many novel techiques to assess the neurological status and create standardized test protocols. One of these techiques is QST(Quantitative Sensory Testing). QST is a specific type of sensory examination, usually done through computerized stimuli of heat, cold or vibration, or specific test equipment. There are many types of QST protocols around the world, and their results can also be expressed as phenotypes through statistics. While there are 3 types of pain phenotypes with the 13 item QST protocol suggested by German Neuropathic Pain Research group(DFNS), all patient groups can be classified differently as well, according to the common findings they express. These different phenotypes are also shown to have different responses to the different pain treatments. Such differences are usually attributed to the different mechanisms and fibers underlying the pathogenesis.

While patients show differences in QST results, evidence for the correlation between these variables and clinical symptoms of the patients are still scarce. Moreover, it is still yet to be known if these differences have a central origin as well as the peripheral mechanisms.

Functional Magnetic Resonance Imaging(fMRI) is a method to evaluate cerebral functions. It is mainly based on the blood flow changes that occur locally in regions that are in function[5]. As a result of the increased blood flow, the oxygen concentration also increases, creating a signal response called BOLD(Blood Oxygen Level Dependent) response. Since different types of pain are conducted through different fibers and pathways, it is also probable that they might show changes in cortical response as well.

In this study, the aim is to find whether QST results are correlated to clinical symptoms and pain properties of the patients, and these changes are related to the changes in the central nervous system

ELIGIBILITY:
Inclusion Criteria:

Adult patients with upper extremity neuropathic pain due to radiculopathy Duration of >1 month Unilateral extremity pain

Exclusion Criteria:

* Severe cognitive impairment
* Unstable systemic comorbidity
* Presence of pacemaker or deep brain stimulation
* Implants that aren't compatible with MRI
* Claustrophobia
* Complete or near complete loss of sensation
* Brain injury or presence intracranial lesions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with upper extremity neuropathic pain due to radiculopathy Duration of >1 month Unilateral extremity pain will be included in the study. Patients will then be stratified according to their total Scores in PainDetect, and neuropathic pain probable or not probable patients will be compared in analyses.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
Functional MRI BOLD responses | Baseline
  In fMRI, patients will first be taking a resting state phase in case of activations. In the block design phase, they will be given tactile stimuli in affected extremity, and then healthy extremity in 3 blocks, followed by pauses in 10 second blocks.

SECONDARY OUTCOMES:
QST(Quantitative Sensory Testing) parameters | Baseline
  QST is planned to be conducted with Case IV system(WR medical Electronics Co. Inc, Maplewood, Minnesota). Their cold threshold, heat threshold, vibration threshold and heat pain threshold will be recorded according to 4,2,1 protocol in both upper extremities. Cold threshold and heat threshold will be expressed as the difference from the skin temperature, expressed as centigrate degrees, through stimuli that are increased or decreased stepwise. For vibration threshold, the stepwise protocol will also be applied, and the results will be recorded as the amplitude of the vibration(micrometers), keeping the frequency constant as 125 Hz. Heat pain threshold will be measured similar to heat sensitivity threshold, and the first painful stimuli and the stimuli which evoked a numeric scale of 5 will be recorded as centigrate degrees(difference from obtained skin temperature).
PainDETECT Questionnaire scores | Baseline
  Patients will be evaluated for the properties of their neuropathic pain with the "PainDetect" inventory, a screening questionnaire. It is composed of questions regarding pain intensity (three numeric rating scales, pain course pattern, a pain drawing reflecting pain radiation, and seven questions addressing somatosensory phenomena which the patient rates on a six-category Likert scale (never-very strongly). A score ranging between 0 and 38, based on the patient's answers in the questionnaire, is calculated. For diagnostic purposes, a validated algorithm has been developed. A painDETECT score ≥19 indicates that a neuropathic pain component is likely, a score of 13-18 is considered uncertain, and a score ≤12 indicates that a neuropathic pain component is unlikely; resulting in three categories of patient pain characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege university school of medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Attal N, Lanteri-Minet M, Laurent B, Fermanian J, Bouhassira D. The specific disease burden of neuropathic pain: results of a French nationwide survey. Pain. 2011 Dec;152(12):2836-2843. doi: 10.1016/j.pain.2011.09.014. Epub 2011 Oct 20. PMID 22019149
- [Background] Magerl W, Krumova EK, Baron R, Tolle T, Treede RD, Maier C. Reference data for quantitative sensory testing (QST): refined stratification for age and a novel method for statistical comparison of group data. Pain. 2010 Dec;151(3):598-605. doi: 10.1016/j.pain.2010.07.026. Epub 2010 Oct 20. PMID 20965658
- [Background] Vollert J, Maier C, Attal N, Bennett DLH, Bouhassira D, Enax-Krumova EK, Finnerup NB, Freynhagen R, Gierthmuhlen J, Haanpaa M, Hansson P, Hullemann P, Jensen TS, Magerl W, Ramirez JD, Rice ASC, Schuh-Hofer S, Segerdahl M, Serra J, Shillo PR, Sindrup S, Tesfaye S, Themistocleous AC, Tolle TR, Treede RD, Baron R. Stratifying patients with peripheral neuropathic pain based on sensory profiles: algorithm and sample size recommendations. Pain. 2017 Aug;158(8):1446-1455. doi: 10.1097/j.pain.0000000000000935. PMID 28595241
- [Background] Holbech JV, Bach FW, Finnerup NB, Jensen TS, Sindrup SH. Pain phenotype as a predictor for drug response in painful polyneuropathy-a retrospective analysis of data from controlled clinical trials. Pain. 2016 Jun;157(6):1305-1313. doi: 10.1097/j.pain.0000000000000563. PMID 27007067
- [Background] Adam A, Dixon AK, Gillard JH, Schaefer-Prokop C, Grainger RG, Allison DJ. Grainger & Allison's Diagnostic Radiology E-Book: Elsevier Health Sciences; 2014.